CLINICAL TRIAL: NCT05753150
Title: Operational Feasibility of Appropriate Plasmodium Vivax Radical Cure With Tafenoquine or Primaquine After Quantitative G6PD Testing in Thailand
Brief Title: Operational Feasibility of Appropriate Plasmodium Vivax Radical Cure After G6PD Testing in Thailand
Acronym: ARCTIC
Status: Completed | Type: Observational
Sponsor: Dr. Prayuth Sudathip (Other Government)
Collaborators: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor-Investigator, Dr. Prayuth Sudathip, Deputy Director, DVBD, Ministry of Health, Thailand
Organization: Ministry of Health, Thailand (Other Government)
Other Study IDs: MMV_TQ_18_01
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Malaria, Vivax; G6PD Deficiency
Keywords: Tafenoquine; Primaquine; G6PD testing; Operational study; Thailand
MeSH Terms: conditions — Malaria, Vivax; Glucosephosphate Dehydrogenase Deficiency | interventions — tafenoquine; Primaquine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Tafenoquine (TQ): Patients aged ≥16 years, G6PD activity ≥ 6.1 U/gHb, not pregnant or breastfeeding, will receive single-dose TQ in addition to chloroquine, the standard blood schizonticidal drug.
  Interventions: Drug: Tafenoquine
- Daily primaquine (PQ) for 14 days: Patients aged ≥16 years, G6PD activity ≥ 4.1 U/gHb, not pregnant or breastfeeding, will receive 14-day PQ in addition to chloroquine, the standard blood schizonticidal drug.
  Interventions: Drug: Primaquine
- Weekly primaquine (PQ) for 8 weeks: Patients aged ≥16 years, G6PD activity ≤ 4.0 U/gHb, not pregnant or breastfeeding, will receive 14-day PQ in addition to chloroquine, the standard blood schizonticidal drug.
  Interventions: Drug: Primaquine

INTERVENTIONS:
Drug: Tafenoquine — Tafenoquine 300 mg (2x150 mg tablets)
  Other Names: Kozenis
  Groups: Tafenoquine (TQ)
Drug: Primaquine — Daily primaquine adjusted by weight (0.25 mg/kg/day for 14 days)
  Groups: Daily primaquine (PQ) for 14 days
Drug: Primaquine — Weekly primaquine adjusted by weight (0.75mg/kg/week for 8 weeks)
  Groups: Weekly primaquine (PQ) for 8 weeks

SUMMARY:
The purpose of this prospective, observational study is to assess the operational feasibility of appropriate radical cure treatment for P. vivax malaria with tafenoquine or primaquine, in patients 16 year and older, after G6PD testing in Thailand. The study will be implemented in a phased manner, in the provinces of Yala and Mae Hong Son. The first phase will be at higher level health facilities (hospitals). An interim analysis will be conducted after 40 patients are enrolled in the study in order to decide whether the study could be extended to lower level HFs. If approved by the Independent Study Oversight Committee, the study will be implemented in lower level HFs (malaria clinics).Higher level HFs will continue to include patients in the study during this 2nd phase.Written informed consent / assent is required from all patients /guardians in the case of minors.

DETAILED DESCRIPTION:
This is a prospective, observational, multi-center, longitudinal study to be conducted in Yala province and Mae Hong Son province in patients with P. vivax malaria.

Since 2020, quantitative G6PD testing has been available for routine use prior to providing PQ radical therapy at district hospitals and malaria clinics in the study provinces, in line with the national guidelines.

Before study start, the relevant staff at all participating sites will be re-trained on the quantitative G6PD test procedure and the radical cure treatment algorithm by the Division of Vector Borne Diseases (DVBD). Standard operating procedures (SOP) for identification of patients with suspected AHA and guidance for initial management and transfer to a referral hospital will be provided.

G6PD tests and TQ will be supplied to Health Facilities (HFs) by the DVBD using the usual supply route for drugs and diagnostics. PQ and other anti-malarial drugs are already available in Thailand.

Within the study period, investigators will prospectively enroll all patients meeting the selection criteria.

Each patient will have to sign an Informed Consent Form (ICF) indicating their consent for participation in the study by being considered for treatment with TQ provided that they have the appropriate G6PD enzyme activity (or treated with PQ, according to the current practice, otherwise) and permitting investigators to use their unidentified data for analysis purposes. Assent from patients <18 years of age, and the parent's or legal guardian's written informed consent must be obtained.

This study will not change the patient/physician relationship, nor influence the investigator's drug prescription or therapeutic management of the patient other than what is specified regarding the algorithm for radical cure treatment of P. vivax malaria with TQ and PQ.

As part of local practice in Yala province and Mae Hong Son province, patients treated for P. vivax infection are asked to return for a follow-up visit on Day 5 (+/- 1 day). This is in addition to the national policy of the first scheduled follow-up visit on Day 14 (+2/- 1 day) for vivax malaria patients. Patient data will be collected by the investigators on each patient visit.

Any suspected case of AHA will be transferred to Yala Referral Hospital, the regional hospital with one board-certified haematologist or to the Mae Hong Son Provincial Hospital. Both hospitals have full services of blood transfusion, renal dialysis, and other life-saving procedures, for further investigation and treatment.

As some patients may not return for the follow-up visits and might develop drug-induced AHA, the study staff at the referral hospitals will regularly screen hospital admission records for malaria patients participating in the study presenting signs of AHA, diagnosed with renal failure, and/or receiving blood transfusion.

The study will be conducted in 2 phases:

* 1st phase (for about 3 months): the study will be implemented in higher level HFs (hospitals). An interim analysis will be conducted after 40 patients (≥16 years old) with P. vivax are enrolled in the study in order to decide whether the study could be extended to lower level HFs. The decision will be made by an Independent Study Oversight Committee (ISOC).
* 2nd phase (approximately 2 months): if approved by the ISOC, the study will be implemented in lower level HFs (malaria clinics).

Higher level HFs will continue to include patients in the study during this 2nd phase.

Final results will be reviewed by the ISOC. It is anticipated that it will take a total of about 11-12 months to complete data collection at the target hospitals and malaria clinics.

ELIGIBILITY:
Inclusion Criteria:

* Thai patient aged ≥16 years at enrolment
* Diagnosed with a mono-species, uncomplicated P. vivax malaria that is parasitologically confirmed through standardized Giemsa microscopy.
* Weighs >35 kg
* Haemoglobin level must be >7gm%
* Less than 24h away from emergency care

Exclusion Criteria:

* Participating in a clinical trial
* Diabetic patients who are (1) being treated with metformin (because of possible increase in the risk of lactic acidosis due to metformin when administered in combination with tafenoquine) (2) G6PD-deficient and being treated with sulfonylureas e.g. Glucotrol, Glynase, Metaglip and Micronase (because of the increased risk of haemolysis in this population).
* Pregnant/lactating women, women with suspected pregnancy.1
* Cases of severe/ complicated malaria

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will be conducted at hospitals and malaria clinics in the provinces of Yala and Mae Hong Son in Thailand.
Sampling Method: Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Appropriate use of TQ based on G6PD activity | 8 months
  Percentage of P. vivax patients aged ≥16 years treated or not with TQ in accordance with the appropriate level of G6PD enzyme activity

SECONDARY OUTCOMES:
Appropriate use of PQ based on G6PD activity | 8 months
  Percentage of P. vivax patients aged ≥16 years treated or not with daily PQ in accordance with the appropriate level of G6PD enzyme activity
Appropriate application of treatment algorithm | 8 months
  Percentage of P. vivax patients who receive TQ or PQ based on the correct application of the treatment algorithm
Reported drug-induced AHA. | 8 months
  Frequency of reported drug-induced AHA.

CONTACTS AND LOCATIONS:
Overall Officials: Chantana Padungtod, M.D., DrPH, Principal Investigator — Director, Dept. Vector Borne Diseases (DVBD); Saowanee Viboonsanti, M.D., Principal Investigator — Director, ODPC Reg. No. 1; Chalermpol Chalermpol, M.D., Principal Investigator — Director, ODPC Reg. No. 12
Locations (9):
- Thailand (9):
  - District Hospital, Mae Sariang, Changwat Mae Hong Son
  - Malaria Clinic, Mae Sariang, Changwat Mae Hong Son
  - District Hospital, Sop Moei, Changwat Mae Hong Son
  - District Hospital, Bannang Sata, Changwat Yala
  - Malaria Clinic, Bannang Sata, Changwat Yala
  - District Hospital, Ka Bang, Changwat Yala
  - Malaria Clinic, Mueang, Changwat Yala
  - District Hospital, Than To, Changwat Yala
  - Malaria Clinic, Than To, Changwat Yala